CLINICAL TRIAL: NCT02006485
Title: A Phase I/Ib Study Evaluating the Efficacy and Safety of Ublituximab, a Third-Generation Anti-CD20 Monoclonal Antibody, in Combination With TGR-1202, a Novel PI3k Delta Inhibitor; and Ibrutinib or Bendamustine, in Patients With B-cell Malignancies.
Brief Title: Ublituximab in Combination With TGR-1202 +/- Ibrutinib or Bendamustine in Patients With B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-103
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — ublituximab; umbralisib; ibrutinib; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ublituximab + TGR-1202 (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions TGR-1202 oral daily dose
  Interventions: Drug: Ublituximab + TGR-1202
- Ublituximab + TGR-1202 + ibrutinib (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions TGR-1202 oral daily dose ibrutinib oral daily dose
  Interventions: Drug: Ublituximab + TGR-1202 + ibrutinib
- Ublituximab + TGR-1202 + bendamustine (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions TGR-1202 oral daily dose Bendamustine at a fixed IV infusion on Days 1 & 2
  Interventions: Drug: Ublituximab + TGR-1202 + bendamustine

INTERVENTIONS:
Drug: Ublituximab + TGR-1202 — Ublituximab IV infusion TGR-1202 oral daily dose
  Arms: Ublituximab + TGR-1202
Drug: Ublituximab + TGR-1202 + ibrutinib — Ublituximab IV infusion TGR-1202 oral daily dose Ibrutinib oral daily dose
  Other Names: Imbruvica
  Arms: Ublituximab + TGR-1202 + ibrutinib
Drug: Ublituximab + TGR-1202 + bendamustine — Ublituximab IV infusion TGR-1202 oral daily dose Bendamustine IV infusion
  Other Names: Treanda
  Arms: Ublituximab + TGR-1202 + bendamustine

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Ublituximab in combination with TGR-1202, with or without ibrutinib or bendamustine, in patients with advanced hematologic malignancies

ELIGIBILITY:
Inclusion Criteria:

* Confirmed B-cell non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), and other B-cell lymphoproliferative disorders as approved by the Medical Monitor or Study Chair
* Refractory to or relapsed after at least 1 prior treatment regimen
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Known hepatitis B virus, hepatitis C virus or HIV infection
* Autologous hematologic stem cell transplant within 3 months of study entry or Allogeneic hematologic stem cell transplant within 12 months
* Primary central nervous system lymphoma or known intracranial involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | 28 days (1 cycle of therapy)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  To assess the overall response rate (ORR) in patients with hematologic malignancies treated with Ublituximab in combination with TGR-1202

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, MD, Study Chair — M.D. Anderson Cancer Center; Susan O'Brien, MD, Study Chair — University of California Irvine Cancer Center
Locations (6):
- United States (6):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Jonesboro, Arkansas
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, Atlanta, Georgia
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Lunning M, Vose J, Nastoupil L, Fowler N, Burger JA, Wierda WG, Schreeder MT, Siddiqi T, Flowers CR, Cohen JB, Sportelli P, Miskin HP, Weiss MS, O'Brien S. Ublituximab and umbralisib in relapsed/refractory B-cell non-Hodgkin lymphoma and chronic lymphocytic leukemia. Blood. 2019 Nov 21;134(21):1811-1820. doi: 10.1182/blood.2019002118. PMID 31558467
- [Derived] Nastoupil LJ, Lunning MA, Vose JM, Schreeder MT, Siddiqi T, Flowers CR, Cohen JB, Burger JA, Wierda WG, O'Brien S, Sportelli P, Miskin HP, Purdom MA, Weiss MS, Fowler NH. Tolerability and activity of ublituximab, umbralisib, and ibrutinib in patients with chronic lymphocytic leukaemia and non-Hodgkin lymphoma: a phase 1 dose escalation and expansion trial. Lancet Haematol. 2019 Feb;6(2):e100-e109. doi: 10.1016/S2352-3026(18)30216-3. PMID 30709431